CLINICAL TRIAL: NCT03832920
Title: Analgesia Nociception Index (ANI) After Unilateral Radical Mastectomy as an Evaluation of Paravertebral Block Failure
Acronym: ANIBPV
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00121-56
Record Dates: First submitted 2019-01-30; First posted 2019-02-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: general anesthesia; paravertebral Block; analgesia nociception index
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analgesia Nociception Index — A monitor of nociception for patients under general anesthesia

SUMMARY:
Paravertebral Block (PVB) combined with general anesthesia (GA) is a conventional pain treatment for breast surgery but sometimes failures can occurs. The efficacy of this block has to be evaluated. Also, for the intra-operative analgesic evaluation of this block, it is necessary to measure intra-operative analgesia index. A monitor of nociception for patients under GA, the PhysiodolorisTM device, offers an index for measuring nociceptive inputs during surgery in anesthetized patients : the ANI index (based on the single R-R interval analysis). The purpose of this observational and prospective study is to assess the variations of this ANI index during breast surgery with or without axillary node dissection with a PVB. This will allow us to quantify the analgesic effect of a PVB during GA for unilateral radical breast surgery with or without axillary node dissection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score (ASA) I or II
* Woman
* Patients aged over 18 years
* BMI between 17 and 30 kg/m2
* Radical mastectomy with or without axillary node dissection.

Exclusion Criteria:

* Preoperative consumption of opioid
* Local Anesthesia allergy
* Local skin inflammation at the puncture area
* Inability to respond to pain assessment using a Numerical Rating Score (NRS)
* Any contra-indication or patient's refusal for regional anesthesia B blocker medication
* Pace maker
* Inability to perform the PVB (at the appreciation of the anesthesiologist)
* Change of surgical procedure other modified radical mastectomy with or without axillary node dissection.
* Patient with a severe side effect or who cannot be controlled by additional therapy will be removed from the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women undergo for a breast surgery with or without axillary node dissection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the ANI index | first minute of the surgical incision
  Assessment of the area under the curve of the variation of the ANI index for the first minute of the surgical incision according to the PVB failure: incomplete or ineffective vs effective. The PVB failure will be evaluate with a cold test on the thoracic levels T2 and T6.

SECONDARY OUTCOMES:
Post Anesthesia Care Unit total dose of morphine will be compare according to the PVB failure or not groups. | Just after surgery (day 0)
  Post Anesthesia Care Unit total dose of morphine will be compare according to the PVB failure or not groups.
Evaluation of pain | Just after surgery (day 0) and the day after surgery (day 1)
  Evaluation of the Numerical Rating Score (NRS) (no pain = 0, worst pain =10): NRS at arrival in the post anesthesia care unit , NRS at leaving of the post anesthesia care unit and at the postoperative day 1. NRS will be compare according to the PVB failure

CONTACTS AND LOCATIONS:
Overall Officials: RAFT JULIEN, MD, Principal Investigator — Institut de Cancérologie de Lorraine (ICL)
Locations (1):
- Institut de Cancérologie de Lorraine (ICL), Vandœuvre-lès-Nancy, France

REFERENCES:
- [Result] Raft J, Lamotte AS, Schohn CH, Fritz C, Richebe P. Analgesia nociception index as a tool to assess the effectiveness of paravertebral block in total mastectomy: a prospective cohort study. Braz J Anesthesiol. 2026 Jan-Feb;76(1):844699. doi: 10.1016/j.bjane.2025.844699. Epub 2025 Nov 7. PMID 41207559
- See also: Related Info — https://doi.org/10.1016/j.bjane.2025.844699